CLINICAL TRIAL: NCT04554498
Title: Toxins Removal and Inflammatory State modulAtion During Online Hemodiafiltration: Comparison of Two Different Dialyzers
Acronym: TRIAD2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Principal Investigator, Gabriele Donati, Principal investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 596/2019/Oss/AOUBo
Record Dates: First submitted 2020-09-05; First posted 2020-09-18 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Hemodialysis Complication; Inflammation; Uremic; Toxemia
MeSH Terms: conditions — Inflammation; Toxemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodiafiltration with ATA filter (Experimental): patients with clinical history of hypersensitivity to polisulfone/poliethersulfone dialysis filters or hypersensitivity to drugs or generic allergens.
  Interventions: Device: 1) high flux hemodiafiltration thrice -weekly during a 24 month follow-up
- Hemodiafiltration with Helixone filter (Active Comparator): no history of hypersensitivity to polisulfone/poliethersulfone dialysis filters is assessed; no history of hypersensitivity to drugs or generic allergens is assessed.
  Interventions: Device: 1) high flux hemodiafiltration thrice -weekly during a 24 month follow-up

INTERVENTIONS:
Device: 1) high flux hemodiafiltration thrice -weekly during a 24 month follow-up — 1. the comparison of the effects of the two membranes on the serum levels of albumin, B2M, CRP, myoglobin, light chains, retinol binding protein, homocysteine, p-cresol, indoxyl sulfate, BPA, alpha-1-microglobulin (A1M), FGF23 (fibroblast growth factor 23), and inflammatory cytokines;
  2. the evaluation of the changes induced by the two filters on lymphocyte subsets, monocyte activation and senescence, and apoptosis rate;
  3. the definition of the impact of the two membranes on the accumulation of AGEs as an index of metabolic and oxidative stress, determined by a non-invasive method based on the measurement of skin autofluorescence through a dedicated device (AGE Reader, DiagnOptics Technologies BV, Groningen, Netherlands).
  Other Names: 2) assessment of uremic toxins, inflammation and effects of patients sera in culture of endothelial cells; 3) Body impedance analysis by means of Electro fluid graph (EFG®, Akern, Pontassieve, Italia); 4) Measurement of AGEs accumulation through skin autofluorescence. (AGE Reader, DiagnOptics Technologies BV)

SUMMARY:
The primary goal of the study is to evaluate in patients on three times a week on-line HDF the efficacy, in terms of toxin removal and modulation of the inflammatory state, of two different dialyzers: Helixone versus Asimmetric cellulose triacetate (ATA).

DETAILED DESCRIPTION:
Patients with end-stage renal disease (ESRD) have a significantly increased cardiovascular mortality rate compared to the general population.

According to the USRDS (United States Renal Data System), in 2017 the prevalence of cardiovascular disease in the United States was 65.8% in patients with chronic kidney disease (CKD), compared to 31.9% of the subjects with stable renal function (https://www.usrds.org/2017/view/v1_04.aspx).

In the natural history of nephropathy, besides the traditional cardiovascular risk factors, an increasingly important role is played by the nontraditional factors related to uremia and dialysis treatment, namely anemia, hyperhomocysteinemia, malnutrition, hyperparathyroidism, electrolyte imbalance, and above all chronic inflammatory state and oxidative stress. The main components of dialysis-related inflammatory response include neutrophil and monocyte activation, cytokine release, oxidative stress with production of free radicals, lipid and protein oxidation, and alterations in blood redox state.

There is much evidence to indicate that ESRD patients, especially those on dialysis, are exposed to increased oxidative and carbonyl stress, that cause chemical modifications of proteins and accumulation of AGEs (advanced glycation end products).

The formation of AGEs occurs through Maillard reaction, a non-enzymatic glycation of peptide amino groups, resulting in protein structural and functional alteration and production of reactive carbonyl species .

Several studies have demonstrated a correlation between the levels of tissue AGEs and the development of various complications, since the accumulation of AGEs constitutes an index of hyperglycemia, oxidative stress and inflammation. The activation and up-regulation of the AGE receptors, including the main one RAGE (AGE Receptor), leads to the initiation of inflammatory cascades involved in the formation of atherosclerotic plaques and endothelial dysfunction, and lastly in the pathogenesis of cardiovascular disease. AGEs are also related to the thickening of the intima-media tunica of the carotid arteries, considered a marker of arteriosclerosis, as clinically confirmed by the close relationship between coronary artery disease and atherosclerotic complications in diabetes and renal failure.

Besides AGEs, a huge pattern of protein-bound toxins and of middle molecular weight uremic toxins are known to contribute to the uremic syndrome in terms of cardiovascular complications, inflammation and fibrosis . Concerning protein-bound uremic toxins, p-cresyl sulfate and indoxyl sulfate have received considerable attention recently. Among middle molecules, B2M, free light chains and FGF23 have been identified as markers of disease progression and mortality in CKD and hemodialysis.

Furthermore, the activation of leukocytes, both in response to the exposure to dialysis membranes and as a consequence of the retrotransportation of substances that promote the expression of cytokines from the dialysate, increases the release of proinflammatory cytokines, such as IL-1β, TNF-α and IL-6.

The biocompatibility and flow properties of the different filters can influence the inflammatory and oxidative response to dialysis and the levels of oxidized molecules. In general, short-term dialysis with high-flow membranes has been shown to decrease plasma levels of oxidized low-density lipoproteins, regardless of the filter material.

Nonetheless, the introduction of high-flux membranes, which increased clearance of middle molecules, appears to be inadequate to improve patient survival, as reported by two major randomized trials, the HEMO study [24] and the MPO study.

The use of on-line HDF, that combines convective and diffusive solute removal, can counterbalance the rapid decrease of middle molecule diffusion obtained with high flux hemodialysis. The integration of diffusion with convection allows a more modest sieving coefficient decrease for middle molecular weight solutes. To date, evidence from four randomized controlled trials on HDF suggests, although not definitely, that HDF with convection volumes >20 L results in better patient outcomes .

Moreover, a correlation of the membrane typology with inflammation and oxidative stress in the medium-long term was found in patients undergoing chronic dialysis treatment. A prospective study in a cohort of 50 patients who started hemodialysis with a high-flux polysulfone membrane (HF80 series, Fresenius Medical Care, St. Wendel, Germany) evaluated the variation of the inflammation and oxidative stress biomarkers. The results showed significantly increased circulating levels of IL-6, C-reactive protein (CRP) and higher carbonylation rate in dialysis patients compared to healthy controls in the first year of observation, and this trend was maintained in the following 12 months.

Successive studies investigated the long-term effects on inflammation and oxidative stress of dialysis with Helixone (Fresenius Medical Care), another type of high-flux polysulfone membrane designed to maximize the clearance of uremic toxins of average molecular weight (> 500 Daltons, Da) compared to conventional high-flux membranes. The introduction of changes as reduced hollow fiber wall thickness (≈35 μm), smaller inner diameter (≈185 μm) and higher average pore size (≈3.3 nm) has improved the clearance of medium molecular weight molecules, including β2-microglobulin (B2M), limiting the passage of larger molecules like albumin, without significant effects on inflammatory parameters .

The features of synthetic membranes related their chemical composition and the asymmetric structure of the fibers make them preferable for new highly-convective therapies, such as high-volume hemodiafiltration (HDF), only partially allowed with cellulose.

However, cellulose triacetate (CTA) and modified cellulose membranes remain the best option for the patients with hypersensitivity reactions to synthetic fibers. Although synthetic membranes, including those based on polysulfone, have a lower risk of hypersensitization than non-biocompatible ones (such as Cuprophane), in some cases adverse reactions have been reported, plausibly due to the contact between the dialyzer itself with plasma proteins and platelets.

Moreover, the choice of polysulfone membranes has been proven to affect the intracellular and serum levels of bisphenol A (BPA, molecular weight 228.3 kDa), a ubiquitous environmental toxicant found in plastic food and beverage containers, as well as in some dialyzers, with several detrimental effects. BPA is considered an endocrine-disrupting chemical that acts mainly as a female hormone: it is associated with reproductive dysfunction, immune abnormality and increased incidence of cancer. Patients on hemodialysis are a high-risk population for BPA overload, because the normal urinary elimination of the conjugated molecule decreases with low renal function. For these reasons, BPA can be thought as a uremic toxin, similarly to p-cresol, and a particular attention should be given to BPA-containing medical devices, including dialysis membranes.

Mas et al. compared BPA-free and BPA-containing dialyzers in 72 patients under on-line HDF, using a prospective 9-month, crossover study design. BPA-free dialyzers determined a greater long-term decrease in BPA levels compared to BPA-containing dialyzers, although at three months the difference was not significant. This may be due to the use of the on-line HDF technique that has been related to lower BPA levels than conventional hemodialysis.

Recently, a new generation filter in asymmetric triacetate (ATA) has been introduced, born from a technology that combines the requirements of synthetic membranes for the possibility of being used with high-volume HDF and the advantages of natural fibers (cellulose) in terms of reduced allergic reactions.

These novel ATA membranes have been demonstrated to achieve satisfactory Kt and convection volume, with good biocompatibility and inflammatory profiles, indicating them as a valuable option for patients allergic to synthetic membranes under HDF treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic renal failure under periodic standard bicarbonate hemodialysis;
* Three times a week dialysis session;
* Residual diuresis <200 mL/day;
* Age >18 years;
* Vascular access for hemodialysis with blood flow >250 mL/minute;
* Need of on-line hemodiafiltration (HDF) for signs of middle molecules intoxication (e.g. B2M >30 mg/L, peripheral neuropathy, cardiovascular comorbidities) or for intradialytic hypotension.

Exclusion Criteria:

* Acute coronary syndrome;
* Acute hemorrage;
* Enrollment in another study protocol;
* Active infection;
* Malignancy;
* Inability to provide written signed consent to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of uremic toxins | 24 months. Blood samples will be drawn at Time 0 (on starting the study when the patients starts HDF treatment), after 1 month, after 3 months, after 6 months, after 12 months, and after 24 months (study end)
  Beta 2 microglobulin (B2M), C-reactive protein (CRP), albumin, myoglobin, light chains, retinol binding protein, homocysteine, p-cresol, indoxyl sulfate, BPA, alpha-2-macroglobulin (A2M), FGF23 (fibroblast growth factor 23)

SECONDARY OUTCOMES:
Measurement of endothelial cells metabolism | 24 months. Blood samples will be drawn at Time 0 (on starting the study when the patients starts HDF treatment), after 1 month, after 3 months, after 6 months, after 12 months, and after 24 months (study end)
  The patients' sera will be incubated with Human Coronary Artery Endothelial Cells (HCAECs), a human cell line isolated from normal coronary arteries. HCAECs are the ideal candidates for the study of endothelial cell functions and metabolism, proving an excellent model system to study all aspects of cardiovascular function and disease
Patients survival | 24 months
  the mortality rate of the patients will be recorded
Body impedance analysis | 24 months.
  Body impedance analysis will be carried out monthly through Electro fluid graph machine
AGEs measurements | 24 months
  AGEs measurements will be carried out monthly through skin autofluorescence
Measurement of inflammatory cytokines | 24 months. Blood samples will be drawn at Time 0 (on starting the study when the patients starts HDF treatment), after 1 month, after 3 months, after 6 months, after 12 months, and after 24 months (study end)
  measurement of interleukin 1 beta (IL-1 β), interleukin 6 (IL-6), interleukin 10 (IL-10),interleukin 12 p 70 (IL-12 (p70)), interleukin 17 (IL -17), tumor necrosis factor alpha (TNF-α) and interferon gamma (IFN-γ)
Measurement of inflammatory cell activation | 24 months. Blood samples will be drawn at Time 0 (on starting the study when the patients starts HDF treatment), after 1 month, after 3 months, after 6 months, after 12 months, and after 24 months (study end)
  Measurement of lymphocyte subsets, monocyte activation and senescence, and apoptosis rate
Infection rate | 24 months
  The number of infections that affected the patients and the rate of hospitalization for infections will be recorded
Cardiovascular diseases | 24 months
  The number of cardiovascular disease that affected the patients and the rate of hospitalization for cardiovascular disease will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano La Manna, Prof, Study Director — StOrsola University Hospital, Bologna, Italy
Locations (1):
- Nephrology Dialysis and Renal Transplantatio Unit, StOrsola University Hospital, Bologna, Italy

REFERENCES:
- [Background] O'Lone E, Viecelli AK, Craig JC, Tong A, Sautenet B, Roy D, Herrington WG, Herzog CA, Jafar T, Jardine M, Krane V, Levin A, Malyszko J, Rocco MV, Strippoli G, Tonelli M, Wang AYM, Wanner C, Zannad F, Winkelmayer WC, Webster AC, Wheeler DC. Cardiovascular Outcomes Reported in Hemodialysis Trials. J Am Coll Cardiol. 2018 Jun 19;71(24):2802-2810. doi: 10.1016/j.jacc.2018.04.012. PMID 29903353
- [Background] Longenecker JC, Coresh J, Powe NR, Levey AS, Fink NE, Martin A, Klag MJ. Traditional cardiovascular disease risk factors in dialysis patients compared with the general population: the CHOICE Study. J Am Soc Nephrol. 2002 Jul;13(7):1918-27. doi: 10.1097/01.asn.0000019641.41496.1e. PMID 12089389
- [Background] Kendrick J, Chonchol MB. Nontraditional risk factors for cardiovascular disease in patients with chronic kidney disease. Nat Clin Pract Nephrol. 2008 Dec;4(12):672-81. doi: 10.1038/ncpneph0954. Epub 2008 Sep 30. PMID 18825155
- [Background] Zoccali C. Cardiovascular risk in uraemic patients-is it fully explained by classical risk factors? Nephrol Dial Transplant. 2000 Apr;15(4):454-7. doi: 10.1093/ndt/15.4.454. No abstract available. PMID 10727537
- [Background] Georgatzakou HT, Tzounakas VL, Kriebardis AG, Velentzas AD, Kokkalis AC, Antonelou MH, Papassideri IS. Short-term effects of hemodiafiltration versus conventional hemodialysis on erythrocyte performance. Can J Physiol Pharmacol. 2018 Mar;96(3):249-257. doi: 10.1139/cjpp-2017-0285. Epub 2017 Aug 30. PMID 28854342
- [Background] Himmelfarb J, McMenamin E, McMonagle E. Plasma aminothiol oxidation in chronic hemodialysis patients. Kidney Int. 2002 Feb;61(2):705-16. doi: 10.1046/j.1523-1755.2002.00151.x. PMID 11849414
- [Background] McIntyre NJ, Fluck RJ, McIntyre CW, Taal MW. Skin autofluorescence and the association with renal and cardiovascular risk factors in chronic kidney disease stage 3. Clin J Am Soc Nephrol. 2011 Oct;6(10):2356-63. doi: 10.2215/CJN.02420311. Epub 2011 Sep 1. PMID 21885790
- [Background] Kimura H, Tanaka K, Kanno M, Watanabe K, Hayashi Y, Asahi K, Suzuki H, Sato K, Sakaue M, Terawaki H, Nakayama M, Miyata T, Watanabe T. Skin autofluorescence predicts cardiovascular mortality in patients on chronic hemodialysis. Ther Apher Dial. 2014 Oct;18(5):461-7. doi: 10.1111/1744-9987.12160. Epub 2014 Jan 24. PMID 24456287
- [Background] Wautier JL, Schmidt AM. Protein glycation: a firm link to endothelial cell dysfunction. Circ Res. 2004 Aug 6;95(3):233-8. doi: 10.1161/01.RES.0000137876.28454.64. PMID 15297385
- [Background] Hangai M, Takebe N, Honma H, Sasaki A, Chida A, Nakano R, Togashi H, Nakagawa R, Oda T, Matsui M, Yashiro S, Nagasawa K, Kajiwara T, Takahashi K, Takahashi Y, Satoh J, Ishigaki Y. Association of Advanced Glycation End Products with coronary Artery Calcification in Japanese Subjects with Type 2 Diabetes as Assessed by Skin Autofluorescence. J Atheroscler Thromb. 2016 Oct 1;23(10):1178-1187. doi: 10.5551/jat.30155. Epub 2016 Mar 10. PMID 26961217
- [Background] Wang CC, Wang YC, Wang GJ, Shen MY, Chang YL, Liou SY, Chen HC, Chang CT. Skin Autofluorescence Is Associated with Endothelial Dysfunction in Uremic Subjects on Hemodialysis. PLoS One. 2016 Jan 25;11(1):e0147771. doi: 10.1371/journal.pone.0147771. eCollection 2016. PMID 26809145
- [Background] Hofmann B, Jacobs K, Navarrete Santos A, Wienke A, Silber RE, Simm A. Relationship between cardiac tissue glycation and skin autofluorescence in patients with coronary artery disease. Diabetes Metab. 2015 Nov;41(5):410-5. doi: 10.1016/j.diabet.2014.12.001. Epub 2014 Dec 29. PMID 25553578
- [Background] Vanholder R, Pletinck A, Schepers E, Glorieux G. Biochemical and Clinical Impact of Organic Uremic Retention Solutes: A Comprehensive Update. Toxins (Basel). 2018 Jan 8;10(1):33. doi: 10.3390/toxins10010033. PMID 29316724
- [Background] Gryp T, Vanholder R, Vaneechoutte M, Glorieux G. p-Cresyl Sulfate. Toxins (Basel). 2017 Jan 29;9(2):52. doi: 10.3390/toxins9020052. PMID 28146081
- [Background] Hung SC, Kuo KL, Wu CC, Tarng DC. Indoxyl Sulfate: A Novel Cardiovascular Risk Factor in Chronic Kidney Disease. J Am Heart Assoc. 2017 Feb 7;6(2):e005022. doi: 10.1161/JAHA.116.005022. No abstract available. PMID 28174171
- [Background] Liabeuf S, Lenglet A, Desjardins L, Neirynck N, Glorieux G, Lemke HD, Vanholder R, Diouf M, Choukroun G, Massy ZA; European Uremic Toxin Work Group (EUTox). Plasma beta-2 microglobulin is associated with cardiovascular disease in uremic patients. Kidney Int. 2012 Dec;82(12):1297-303. doi: 10.1038/ki.2012.301. Epub 2012 Aug 15. PMID 22895515
- [Background] Desjardins L, Liabeuf S, Lenglet A, Lemke HD, Vanholder R, Choukroun G, Massy ZA; European Uremic Toxin (EUTox) Work Group. Association between free light chain levels, and disease progression and mortality in chronic kidney disease. Toxins (Basel). 2013 Nov 8;5(11):2058-73. doi: 10.3390/toxins5112058. PMID 24217396
- [Background] Gutierrez OM, Mannstadt M, Isakova T, Rauh-Hain JA, Tamez H, Shah A, Smith K, Lee H, Thadhani R, Juppner H, Wolf M. Fibroblast growth factor 23 and mortality among patients undergoing hemodialysis. N Engl J Med. 2008 Aug 7;359(6):584-92. doi: 10.1056/NEJMoa0706130. PMID 18687639
- [Background] Menegatti E, Rossi D, Chiara M, Alpa M, Sena LM, Roccatello D. Cytokine release pathway in mononuclear cells stimulated in vitro by dialysis membranes. Am J Nephrol. 2002 Sep-Dec;22(5-6):509-14. doi: 10.1159/000065288. PMID 12381952
- [Background] Memoli B, Postiglione L, Cianciaruso B, Bisesti V, Cimmaruta C, Marzano L, Minutolo R, Cuomo V, Guida B, Andreucci M, Rossi G. Role of different dialysis membranes in the release of interleukin-6-soluble receptor in uremic patients. Kidney Int. 2000 Jul;58(1):417-24. doi: 10.1046/j.1523-1755.2000.00181.x. PMID 10886590
- [Background] Walker RJ, Sutherland WH, De Jong SA. Effect of changing from a cellulose acetate to a polysulphone dialysis membrane on protein oxidation and inflammation markers. Clin Nephrol. 2004 Mar;61(3):198-206. doi: 10.5414/cnp61198. PMID 15077871
- [Background] Furuta M, Kuragano T, Kida A, Kitamura R, Nanami M, Otaki Y, Nonoguchi H, Matsumoto A, Nakanishi T. A crossover study of the acrylonitrile-co-methallyl sulfonate and polysulfone membranes for elderly hemodialysis patients: the effect on hemodynamic, nutritional, and inflammatory conditions. ASAIO J. 2011 Jul-Aug;57(4):293-9. doi: 10.1097/MAT.0b013e31821796f1. PMID 21499075